CLINICAL TRIAL: NCT00427245
Title: Ovarian Protection Trial In Premenopausal Breast Cancer Patients [OPTION]
Brief Title: Goserelin in Preventing Early Menopause in Premenopausal Women Undergoing Chemotherapy for Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anglo Celtic Cooperative Oncology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CRUK-OPTION; CDR0000526368 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2004-000133-11; CRUK-BR0402; ISRCTN84856516; EU-20680
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer; Infertility; Menopausal Symptoms
Keywords: menopausal symptoms; infertility; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Infertility | interventions — Cyclophosphamide; Goserelin; Chemotherapy, Adjuvant; Therapeutics; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: goserelin acetate
Procedure: adjuvant therapy
Procedure: fertility assessment and management
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Goserelin may help prevent early menopause in patients undergoing chemotherapy for breast cancer. It is not yet known whether goserelin is effective in preventing early menopause in women undergoing chemotherapy for breast cancer.

PURPOSE: This randomized phase III trial is studying goserelin to see how well it works compared with no goserelin in preventing early menopause in premenopausal women undergoing chemotherapy for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of premature ovarian failure after chemotherapy in premenopausal women with stage I-III breast cancer treated with goserelin vs no goserelin .

Secondary

* Compare the quality of life of patients treated with these regimens.
* Compare menopausal symptoms in patients treated with these regimens.
* Compare bone mineral density loss in patients treated with these regimens.
* Compare hormone levels in patients treated with these regimens.
* Compare menstruation in patients treated with these regimens.
* Compare the incidence of pregnancy in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, prospective, parallel group, multicenter study. Patients are stratified according to age (≤ 40 years vs > 40 years) and participating center. Patients are randomized to 1 of 2 treatment arms.

Arm I (chemotherapy alone): Patients receive neoadjuvant or adjuvant cyclophosphamide- and/or anthracycline-containing chemotherapy. Treatment continues for 6-8 courses in the absence of disease progression or unacceptable toxicity.

Arm II (chemotherapy plus goserelin for ovarian function suppression): Patients receive neoadjuvant or adjuvant chemotherapy as in arm I. Patients also receive goserelin subcutaneously every 3-4 weeks beginning 1-3 weeks before the start of chemotherapy. Treatment with goserelin repeats every 3-4 weeks until completion of chemotherapy.

Quality of life is assessed at baseline, at 3, 6, 12, 18, and 24 months, and then annually for up to 5 years.

After completion of study therapy, patients are followed periodically for 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stages I-IIIB with node-positive or -negative disease (N0-2)
  * Operable disease
* Must meet 1 of the following criteria:

  * Has undergone mastectomy or breast-conserving surgery with complete excision of primary tumor within the past 8 weeks
  * Scheduled to receive neoadjuvant chemotherapy
* No metastatic breast cancer, including supraclavicular fossa metastases
* Hormone receptor status meeting 1 of the following criteria:

  * Estrogen receptor (ER) and progesterone receptor poor or negative AND not a candidate for adjuvant endocrine therapy
  * ER positive AND no requirement for ovarian suppression as a necessary part of treatment

PATIENT CHARACTERISTICS:

* Female
* Premenopausal with regular menses in the 12 months preceding surgery
* No other prior or concurrent invasive malignancy except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Suitable fitness status for chemotherapy
* Adequate hepatic, renal, and bone marrow function
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or endocrine therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Rate of premature menopause, defined as cessation of menses during a course of chemotherapy with no recovery for at least 12 months

SECONDARY OUTCOMES:
Incidence of menopausal symptoms
Quality of life
Bone mineral density loss as measured by dual energy X-ray absorptiometry scans at 12, 24, and 36 months and by serum biomarkers
Hormone levels (including follicle-stimulating hormone, luteinizing hormone, beta-inhibin, and estradiol) as measured after course 3, after course 6 or 8 (depending on chemotherapy regimen), at 9 and 12 months, and then annually for up to 5 years
Menstruation history as measured by patient menstrual diary for 24 months from the start of chemotherapy
Incidence of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Robert C.F. Leonard, MD, BS, MB, Study Chair — Charing Cross Hospital
Locations (66):
- United Kingdom (66):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Frenchay Hospital, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Halton Hospital, Cheshire, England
  - Essex County Hospital, Colchester, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - UCL Cancer Institute, Hampstead, London, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - King George Hospital, Ilford, Essex, England
  - Ipswich Hospital, Ipswich, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Yorkshire Regional Clinical Trials & Research Unit, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Whipps Cross Hospital, London, England
  - Newham University Hospital, London, England
  - Homerton University Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Whittington Hospital, London, England
  - Guy's Hospital, London, England
  - St. George's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Luton and Dunstable Hospital, Luton-Bedfordshire, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - North Manchester General Hospital - Penine Actute Hospitals Trust, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Oldchurch Hospital, Romford, England
  - Salisbury District Hospital, Salisbury, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Kent and Sussex Hospital, Tunbridge Wells, Kent, England
  - Warrington Hospital NHS Trust, Warrington, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - New Cross Hospital, Wolverhampton, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Queen Margaret Hospital - Dunfermline, Dunfermline, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - Royal Glamorgan Hospital, Lhantrisant, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales